CLINICAL TRIAL: NCT06865911
Title: Cold Versus Warm Tumescent Solution in Arm Liposculpture: A Double-blind Clinical Study.
Brief Title: Cold Versus Warm Tumescent Solution in Arm Liposculpture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eternal Beauty SAS (Other)
Responsible Party: Principal Investigator, Laura Cristina Cala Uribe, Plastic Surgeon, Eternal Beauty SAS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CP_ArmCOLD001; Cold Arms (Other: Eternal Beauty SAS)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Arm Pain; Arm Aesthetics; Liposuction; Safety of Intervention
Keywords: Tumescent solution; Arm liposculpture; Cold anesthesia; VASER-assisted lipoplasty; Liposuction outcomes
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prevention of excessive edema, pain and ecchymosis after liposculpture with the use of cold tumescent solution.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold tumescent solution (Experimental): 1. Cold Tumescent Solution Group: Infiltration of tumescent solution at 4°C. Composition of tumescent solution: 1000 ml of Ringer's lactate + 7 ml of 2% Lidocaine without Epinephrine + 1 mg of Epinephrine + 250 mg of Tranexamic Acid.
  Interventions: Other: Cold crystalloid infusions, 0.9%NaCl or Ringer's; Procedure: Liposuction of the arms
- Warm tumescent solution (Placebo Comparator): 2. Warm Tumescent Solution Group: Infiltration of tumescent solution at room temperature. Composition of tumescent solution: 1000 ml of Ringer's lactate + 7 ml of 2% Lidocaine without Epinephrine + 1 mg of Epinephrine + 250 mg of Tranexamic Acid.
  Interventions: Other: Warm saline; Procedure: Liposuction of the arms

INTERVENTIONS:
Other: Cold crystalloid infusions, 0.9%NaCl or Ringer's — Infiltration of cold tumescent solution at 4 C for lipoplasty.
  Other Names: Tumescent solution
  Arms: Cold tumescent solution
Other: Warm saline — Infiltration of warm tumescent solution at body temperature for lipoplasty.
  Other Names: Warm tumescent solution
  Arms: Warm tumescent solution
Procedure: Liposuction of the arms — Infiltration of tumescent solution in both arms, VASER fat emulsification then power-assisted liposuction of the arms.

SUMMARY:
The goal of this clinical trial is to evaluate whether the temperature of tumescent solution (cold vs. warm) affects postoperative outcomes in adults undergoing arm liposculpture. The study includes men and women aged 18-60 years with certain body complexity, however no obese patients are allowed to enter the study. All patients are undergoing bilateral arm liposculpture as part of body contouring procedures.

The main questions it aims to answer are:

* Does using a cold tumescent solution reduce postoperative bruising compared to a warm solution?
* Does a cold tumescent solution reduce postoperative inflammation compared to a warm solution?
* How does solution temperature affect the quality of fat samples collected during liposuction?

Researchers will compare the cold tumescent solution group to the warm tumescent solution group to determine whether a lower temperature provides benefits in terms of reduced bruising, inflammation, and improved fat quality.

Participants will:

* Receive either a cold (4°C) or warm (room temperature) tumescent solution in each arm before liposuction.
* Undergo fat emulsification with VASER technology.
* Have one arm treated with Power-Assisted Liposuction (PAL) and the other with Conventional Suction-Assisted Liposuction (SAL).
* Have liposuction fat samples collected for analysis of fat content, blood content, and overall fat quality.
* Be monitored for bruising and inflammation on Days 1, 3, and 7 using an image analyzing software and arm circumference measurements.
* Complete a satisfaction survey 30 days after surgery.

Safety considerations include monitoring core temperature and using external warming devices if needed to prevent hypothermia.

DETAILED DESCRIPTION:
Study Objective:

To compare the effects of cold (4°C) and warm tumescent solutions in arm liposculpture on postoperative outcomes, specifically in terms of inflammation, bruising, and fat emulsification using different liposuction techniques.

Study Design

* Type: Interventional (Clinical Trial)
* Allocation: Randomized
* Intervention Model: Parallel Assignment
* Masking: Double-blind (Participants and Surgeon)
* Primary Purpose: Prevention of complications

Population: Adults aged 18-60 years scheduled for bilateral arm liposculpture together with other body contouring procedures.

Interventions

1. Cold Tumescent Solution Group (Intervention arm)

   o Infiltration of tumescent solution at 4°C.
2. Warm Tumescent Solution Group (Control arm) o Infiltration of standard tumescent solution (room temperature).

Tumescent Solution Composition (for both groups):

* 7 cc of 2% Lidocaine without Epinephrine.
* 1 mg of Epinephrine.
* 250 mg of Tranexamic Acid.

Procedure Outline

1. Infiltration Phase: Each arm is infiltrated with its respective tumescent solution (cold or warm). Allow a 15-minute diffusion period for the tumescent solution to take effect.
2. VASER Emulsification: Apply VASER technology to both arms at 50% power for fat emulsification.
3. Liposuction Techniques: Arm A: Liposculpture performed using Power-Assisted Liposuction (PAL). Arm B: Liposculpture performed using Conventional Suction-Assisted Liposuction (SAL).
4. Fat is collected separately for each arm and stored in individual containers.
5. Sample Collection for Analysis:

   * Collect a lipocrit sample in a 10 ml syringe from each arm.
   * Send the samples to pathology for analysis of fat content, blood content, and overall quality of the liposuction sample.

Primary Outcome Measures

1. Postoperative Bruising: Assessed using ImageJ software to quantify areas of bruising at Days 1, 3, and 7 postoperative.
2. Inflammation: Measured via arm circumference on Days 1, 3, and 7.
3. Quality of Fat Samples: Pathological evaluation of fat and blood content from the lipocrit samples.

Secondary Outcome Measures

1. Patient Satisfaction: Surveys conducted 30 days post-procedure.
2. Complication Rates: Hematoma, seroma, and infection rates evaluated within 30 days post-op.

Safety Considerations:

Surgeons must be cautious when using cold tumescent solutions due to the risk of hypothermia, particularly during extended procedures. Continuous core temperature monitoring and the use of external warming devices are recommended to mitigate the risks of lowering core temperature.

Timeline:

* Start Date: January 2023
* Primary Completion Date: December 2023
* Study Completion Date: June 2024

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years.
* Body mass index between 18 and 30.
* Patients scheduled for bilateral arm liposculpture together with other body contouring procedures.
* Able to provide informed consent.

Exclusion Criteria:

* History of coagulopathies.
* ASA > II.
* Allergies to tumescent solution components (epinephrine, lidocaine).
* Pregnant or lactating individuals.
* Previous surgeries on the arms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Ecchymosis | 7 days
  1. Postoperative Bruising: Assessed using ImageJ software to quantify areas of bruising at Days 1, 3, and 7 postoperative.
Edema/inflammation | 7 days
  2. Inflammation: Measured via arm circumference on Days 1, 3, and 7.
Pain score | 7 days
  3. Postoperative pain: Scoring system using the visual analogue scale. From 1 to 10 at each time point: immediately after surgery, 1 ,3 and 7 days postoperative.

SECONDARY OUTCOMES:
Lipocrit evaluation | 6 hours
  4. Quality of Fat Samples: Pathological evaluation of fat and blood content from the lipocrit samples.
Patient satisfaction | 30 days
  1. Patient Satisfaction: Surveys conducted 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio E Perez Pachon, MD, Study Director — Total Definer
Locations (1):
- Dhara Clinic, Bogota DC, Bogota DC, Colombia

IPD SHARING:
Plan to Share IPD: No
There is patient information that cannot be disclosed due to patient preferences.

REFERENCES:
- [Background] Hoyos AE, Perez Pachon ME, Benavides JE, Eljaiek A, Borras Osorio M, Ramirez B. Effects of Optimal Temperature Control in Body Contouring Surgery: A Nonrandomized Controlled Clinical Trial. Aesthet Surg J. 2024 Oct 15;44(11):NP790-NP797. doi: 10.1093/asj/sjae142. PMID 38953184
- [Background] Hoyos A, Perez M. Arm dynamic definition by liposculpture and fat grafting. Aesthet Surg J. 2012 Nov;32(8):974-87. doi: 10.1177/1090820X12461498. PMID 23110928
- [Background] Cala Uribe LC, Perez Pachon ME, Babaitis R, Zannin Ferrero A, Aljure Diaz MF. Variable Energy and Ultrasound-based Liposculpture of the Arms: Multicenter and Multidevice Study. Plast Reconstr Surg Glob Open. 2024 Mar 19;12(3):e5649. doi: 10.1097/GOX.0000000000005649. eCollection 2024 Mar. PMID 38948160
- [Background] Cala Uribe LC, Perez Pachon ME, Zannin Ferrero A, Neri Morales C, Silva Gutierrez J, Manrique Cruz AD, Maza MF, Acero Mondragon EJ, Celis Regalado LG. Effects of Bipolar Radiofrequency on Collagen Synthesis from Patients with Brachial Ptosis. Plast Reconstr Surg Glob Open. 2023 Apr 13;11(4):e4924. doi: 10.1097/GOX.0000000000004924. eCollection 2023 Apr. PMID 37063507